CLINICAL TRIAL: NCT00585728
Title: CT Virtual Proctoscopy for Staging and Volume Assessment for Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007-0134 (CC07206); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); 2007-0134 (Other: Institutional Review Board)
Record Dates: First submitted 2007-12-21; First posted 2008-01-03 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2011-08

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): CT virtual proctoscopy
  Interventions: Procedure: CT Virtual Proctoscopy (CTVP)

INTERVENTIONS:
Procedure: CT Virtual Proctoscopy (CTVP) — CTVP done prior to initiation of therapy and a couple of weeks before patient has surgery.

SUMMARY:
The purpose of this study is to see how CT virtual proctoscopy compares to an ultrasound exam of the rectal area in determining the stage of rectal cancer for people recently diagnosed with rectal cancer. This study will also compare tumor volume before and after neoadjuvant therapy using CT virtual proctoscopy, with the ultrasound exam as a comparison. Neoadjuvant therapy consists of chemotherapy and radiation therapy. Neoadjuvant chemoradiation therapy is done before surgery to reduce the size of tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with adenocarcinoma of the rectum, who have not started their neoadjuvant treatment yet.

Exclusion Criteria:

* Patients who have started their neoadjuvant therapy already

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The utility of CT virtual proctoscopy (CTVP) for evaluation of rectal cancer. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles P Heise, M.D., Principal Investigator — UW Hospital & Clinics, Department of Surgery
Locations (1):
- University of Wisconsin Hospital & Clinics, Madison, Wisconsin, United States